CLINICAL TRIAL: NCT06518109
Title: Caregiver's Burden and Their Relationship to Physical Activity, Exercise Self-Efficacy, Perceived Exercise Benefits and Barriers in Caregivers of Children With Autism Spectrum Disorder
Brief Title: Caregivers of Children With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Güllü Aydın Yağcıoğlu, Assistant Professor, Gulhane School of Medicine
Other Study IDs: CCA
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Caregiver Burden; Exercise; Physical Activity
MeSH Terms: conditions — Autism Spectrum Disorder; Caregiver Burden; Motor Activity | interventions — Zarit Caregiver Burden Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Zarit Caregiver Burden Scale — The Zarit Caregiver Burden Scale (ZCBS) is a widely used instrument for assessing the burden experienced by caregivers of individuals requiring long-term care. It consists of 22 items and the total score ranges from 0 to 88 (low/no burden to severe burden)

SUMMARY:
This study aims to examine the relationship between caregiving burden and physical activity, exercise self-efficacy, and perceived exercise benefits and barriers in caregivers of Caregivers of children with autism spectrum disorder (CwASD).The study population consisted of primary caregivers of a CwASD for at least 1 year. Caregiving burden was assessed using the Zarit Caregiver Burden Scale, physical activity using the International Physical Activity Questionnaire-Short form (IPAQ-SF), exercise self-efficacy using the Exercise Self-Efficacy Scale, and perceived exercise benefit using the Exercise Benefits/Barriers Scale. The relationship between caregiver burden and other parameters was analysed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Caring for a CwASD for at least 1 year,
* The child with autism is 18 years old or younger,
* being an informal carer,
* The caregiver is the person with primary responsibility for the care of the CwASD in the family.

Exclusion Criteria:

* People over the age of 65,
* Those without a diagnosed chronic physical condition leading to disability,
* Those caring for more than one CwASD, another disabled person, an older adult or someone needing care

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population were being over 18 years of age, caring for a CwASD for at least 1 year, the child with autism being 18 years of age or younger, being an informal caregiver, and the caregiver being the person with primary responsibility for caring for the CwASD in the family.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
The Zarit Caregiver Burden Scale | 10 minutes
  The Zarit Caregiver Burden Scale (ZCBS) is a widely used instrument for assessing the burden experienced by caregivers of individuals requiring long-term care. It consists of 22 items and the total score ranges from 0 to 88 (low/no burden to severe burden)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided